CLINICAL TRIAL: NCT06944054
Title: Evaluation of the Effect of the Time the Stabilizer Tapes Stay on the Skin on Skin Damage in Newborns
Brief Title: Evaluation of the Effect of Duration of Stabilising Tapes on Skin Damage in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-HF-KK-01
Record Dates: First submitted 2025-01-13; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-12

CONDITIONS: Newborns
Keywords: Skin Damage; Epidermis; Stabilization Tapes; Newborn

STUDY DESIGN:
Intervention Model Description: Participants were divided into experimental and control groups. In the experimental group, the fixative tapes were changed every 2 hours, and in the control group, the clinical routine was applied and changed every 4 hours.
Masking Description: In the study, participant and researcher blinding could not be performed because the researcher was involved in the application and the method applied to the parents of the participants was explained verbally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 hourly interval stabiliser band change group (Experimental): Every 2 hours, the heat probes were replaced. Hypoallergenic patches were removed with a silicone-based spray used in the clinic. The application continued for 24 hours. In total, 12 heat probe displacements were made to different points in the abdominal, chest or lower extremity region. Heat probe stabilising tapes were attached to different points in a clockwise direction. At the end of 24 hours, the skin conditions of the newborns were re-evaluated with scales and recorded. This application continued for 3 days.
  Interventions: Other: Group 1
- 4 hourly interval stabiliser band change group (No Intervention): Hypoallergenic patches were removed with a silicone-based spray used in the clinic. The application continued for 24 hours. A total of 6 heat probe displacements were applied to different points in the abdomen, chest or lower extremities at 4-hour intervals. Heat probe fixation bands were attached clockwise to different points. At the end of 24 hours, the skin condition of the newborns was evaluated with scales. This application continued for 3 days.

INTERVENTIONS:
Other: Group 1 — Every 2 hours, the heat probes were replaced. Hypoallergenic patches were removed with a silicone-based spray used in the clinic. The application continued for 24 hours. In total, 12 heat probe displacements were made to different points in the abdominal, chest or lower extremity region. Heat probe stabilising tapes were attached to different points in a clockwise direction. At the end of 24 hours, the skin conditions of the newborns were re-evaluated with scales and recorded. This application continued for 3 days.
  Arms: 2 hourly interval stabiliser band change group

SUMMARY:
The research was conducted to evaluate the relationship between the duration of the fixing tapes of the probes attached to the chest, abdominal and lower extremity regions of newborns for temperature monitoring and skin damage.

DETAILED DESCRIPTION:
Aim: The research was conducted to evaluate the relationship between the duration of the fixing tapes of the probes attached to the chest, abdominal and lower extremity regions of newborns for temperature monitoring and skin damage.

Materials and Methods: The research was conducted in a randomized controlled experimental design between August 2023 and December 2023. The 37th-40th year is being treated in the Neonatal Intensive Care Unit of Gynecology Training and Research Hospital. It was done with 60 newborns between weeks. Newborns were assigned to the experimental group (n = 30) and control group (n = 30) by simple randomization. In the experimental group, the duration of the fixative tapes to stay on the skin was 2 hours, and in the control group, the duration of the fixative tapes to stay on the skin was 4 hours, which is applied in the clinical routine. Stabilizer tapes were adhered to three different areas on the skin and changed clockwise. Data were collected using the Newborn Information Form, Newborn Skin Condition Assessment Scale (NSCS) and Newborn Skin Risk Assessment Scale (NSRAS). Descriptive statistics, repeated measures ANOVA, Pearson Correlation test and Pearson Chi Square test statistics were used in data analysis. p<0.05 level was considered statistically significant.

Key Words: Newborn, Skin Damage, Epidermis, Stabilization Tapes, Newborn Nurse

ELIGIBILITY:
Inclusion Criteria:

* Newborns between 37th and 40th week
* Use of a temperature monitoring probe
* Parents volunteering their infants to participate in the study and signing the consent form

Exclusion Criteria:

* Presence of conditions that may make skin condition assessment difficult (presence of any laceration, fracture or genetic dermatological disease that disrupts skin integrity, congenital skin damage, hydrops, anomalies of the anterior abdominal wall, scleroderma)
* Parents not volunteering for the study

Ages: 37 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Skin Condition Assessment Scale (NSCS) | 3 days
  The NSCS is a 3-point Likert-type scale that evaluates dryness, redness, peeling and deterioration of the skin. Evaluation of the scale score: each criterion was scored with 1 being the best and 3 being the worst. A maximum of 9 and a minimum of 3 points can be scored in the total score. A score of 9 indicates a poor skin score, while a score of 3 indicates a good skin score. An increase in the scale score means that the skin condition is poor.
Neonatal Skin Risk Assessment Scale | 3 days
  These are general physical condition, mental state, mobility, activity, nutrition, humidity. Each parameter in the scale is scored from 1 to 4. The score that can be obtained from the scale varies between 6 and 24. A high score on the scale indicates an increased risk of skin integrity disruption in the newborn, while a low score means that the risk of skin integrity disruption is low. was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlik Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No